CLINICAL TRIAL: NCT07388303
Title: The Relationship Between Perceived Manual Ability and Functional Measurements in Patients With Hand-Forearm Injuries
Brief Title: Perceived Ability and Hand Function
Status: Recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-125116
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hand Injuries; Forearm Injuries
Keywords: hand forearm injuries; perceived manual ability; functional measurements
MeSH Terms: conditions — Hand Injuries; Forearm Injuries | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated conservatively or surgically in the orthopedics clinic due to hand-forearm injuries
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — The Modified Hand Injury Severity Score is used to determine the severity level of patients' injuries. At the 6th and 12th weeks following the injury or surgery, patients are administered the Manual Ability Measure-36 questionnaire, and the Jebsen-Taylor Hand Function Test and Nine-Hole Peg Test are performed. Additionally, the grip strength of the subjects is evaluated at the 12th week.

SUMMARY:
Patient-reported outcome measures, which are subjective by nature, need to be correlated with clinician-administered professional measurements as a further step toward expanding their clinical utility. Therefore, this study aimed to investigate the relationship between perceived manual dexterity and functional measurements in patients with hand-forearm injuries.

ELIGIBILITY:
Inclusion Criteria:

* Having sustained a hand and/or forearm injury and/or having undergone surgery related to this injury.
* Being voluntary to participate in the study.

Exclusion Criteria:

* Patients with concomitant central nervous system involvement.
* Patients with a history of previous injury to the same extremity.
* Patients with rheumatological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated conservatively or surgically in the orthopedics clinic due to hand-forearm injuries
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The Modified Hand Injury Severity Score | At baseline
  It is a four-component scoring system developed to determine the severity of hand and forearm injuries: integumentary (skin and nail), skeletal (bone and ligament), motor (tendon), and neurovascular (nerve and vascular). The total score is obtained by summing the scores of all components and is classified into four categories: minor (<20), moderate (21-50), severe (51-100), and major (>101) injury.
Manual Ability Measure-36 | At the 6th and 12th weeks following injury or surgery
  It is a self-report questionnaire specifically developed to measure hand dexterity. It is an outcome measure that reflects patients' perceived functional hand use or their ability to perform activities of daily living. Higher scores indicate higher levels of function.
The Jebsen-Taylor Hand Function Test | At the 6th and 12th weeks following injury or surgery
  It consists of seven subtests: writing, turning over cards, picking up small common objects, simulated feeding, stacking checkers, moving light objects, and moving heavy objects.
The Nine-Hole Peg Test | At the 6th and 12th weeks following injury or surgery
  It is a simple, rapid, and manual dexterity test with proven validity and reliability. It is particularly sensitive to changes in upper extremity performance.
Gross and fine grip strength | At the 6th and 12th weeks following injury or surgery
  These measurements are performed according to the procedure recommended by the American Society of Hand Therapists.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Eraslan, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rallon, C. R., & Chen, C. C. (2008). Relationship between performance-based and self-reported assessment of hand function. American Journal of Occupational Therapy, 62(5), 574-579.
- [Background] Chen, C. C., & Bode, R. K. (2010). Psychometric validation of the Manual Ability Measure-36 (MAM-36) in patients with neurologic and musculoskeletal disorders. Archives of physical medicine and rehabilitation, 91(3), 414-420.